CLINICAL TRIAL: NCT03167385
Title: The Effectiveness and Safety of Apatinib Mesylate in Locally Advanced/Metastatic Differentiated Thyroid Carcinoma: a Phase 2 Trial.
Brief Title: Phase 2 Trial of Apatinib Mesylate in Locally Advanced/Metastatic Differentiated Thyroid Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBT001
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-03

CONDITIONS: Differentiated Thyroid Carcinoma
Keywords: locally advanced differentiated thyroid carcinoma; radioiodine refractory thyroid carcinoma
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experitmental (Experimental): Continuous oral intake of Apatinib Mesylate (500mg), once a day, until progression of disease or severe adverse effect.
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — oral intake of Apatinib Mesylate 500mg once a day until progression of diesase or severe adverse effect
  Other Names: YN968D1

SUMMARY:
This is a non-randomized, phase II, open label study of Apatinib Mesylate in patients with with locally advanced or metastatic differentiated thyroid carcinoma (DTC). The purpose of this study is to evaluate the efficacy and safety of apatinib in patients with locally advanced or metastatic differentiated thyroid carcinoma.

DETAILED DESCRIPTION:
At present, multiple anti-angiogenesis drugs for thyroid cancer of clinical research are ongoing worldwide, and most of which achieved fairly good therapeutic effect. To date, sorafenib has been approved for the treatment of radioactive iodine refractory DTC. Apatinib is a highly selective VEGFR2 inhibitor that reduces the angiogenesis of tumor efficiently, and had been proven to be effective in many solid tumors. In this study, the investigators aim to further explore the efficacy and safety of apatinib in locally advanced or metastatic differentiated thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Histopathology confirmed locally advanced or metastatic differentiated thyroid carcinoma, with measurable lesions (RECIST 1.1).
3. Age:18-75 years, ECOG（Eastern Cooperative Oncology Group） Score:0-2, Expected survival period ≥ 3 months.
4. Patients with disease progression which was confirmed by imaging in 18 months, and meet any one of the following four:

   1. The tumor invades important organs, and cannot be resectted completely, the remnant thyroid tissue is extensive and not suitable for further iodine treatment.
   2. Lesions have no iodine affinity.
   3. The cumulative dose of RAI (radioactive iodine) ≥ 600mCi or 22GBq.
   4. Patients with disease progression confirmed by radiological examination within 18 months of last RAI.
5. Patients general condition meeting the following:

   Haemoglobin (HBG) ≥ 90 g/L, neutrophil count (ANC) ≥ 1.5×109/L, platelet count (PLT) ≥ 80×109/L, total bilirubin (TBIL)< 1.5×ULN (upper limit of normal), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5×ULN (ALT and AST < 5×ULN if have liver metastasis), SCr (serum creatinine) <1.5×ULN, left ventricular ejection fraction ≥ 50% of normal.
6. Past history of less than one kind of tyrosine kinase inhibitor.
7. Pregnancy test (serum or urine) has to be performed in woman of childbearing age within 7 days before enrolment and the test result must be negative. Patients enrolled should take appropriate contraceptive measures during the study until the 6th month post the last administration of study drug. For male participants, (previous surgical sterilization accepted), agreement to take appropriate methods of contraception during the study until the 6th month post the last administration of study drug is required.

Exclusion Criteria:

1. Patients with past apatinib treatment or have received two or more small molecular TKI (Tyrosine Kinase Inhibitor) drugs.
2. Patients accepted external beam radiation therapy or iodine - 131 therapy in recent three months, or patients plan to receive the other systemic anti-tumor treatment during the study.
3. Patient with history of another malignant disease within past 5 years, cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor are spared.
4. Patients without unrelieved toxicity reaction above CTCAE grade, neurotoxicity and hair loss due to oxaliplatin are spared.
5. Preconditions that impair successful oral medication intake (such as inability to swallow, chronic diarrhea).
6. Patients with pleural effusion or ascites that lead to respiratory syndrome (above CTCAE grade 2).
7. Patients with severe systemic diseases that might impair cardiac function, et al.
8. Patients accepted major surgery、incision biopsy or obvious traumatic injury in 28 days before the study.
9. Patients with physical signs or medical history of bleeding.
10. Patients with thromboembolism event in 6 months.
11. Patients with history of aneurysm.
12. Patients with epilepsy which needs medication.
13. Patients with history of psychiatric drug abuse or have a mental disorder.
14. Patients with history of disease in peripheral nervous system, muscle strength under level 3.
15. Attended other antitumor drug clinical trials or other ongoing clinical subjects within 4 weeks.
16. According to the researcher's judgment, there is other possible serious condition that endanger the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
disease control rate | within two weeks of drug administration
  percentage of patients who have achieved complete response, partial response and stable disease to overall therapeutic intervention patients

SECONDARY OUTCOMES:
progression free survival | 2 years
  time that passes from the day the participants received the apatinib and the date on which disease progresses or the date on which the patient dies, from any cause.
overall survival | 2 years
  percentage of patients who are alive after a certain time period after they were treated
objective response rate | 2 weeks
  percentage of patients who have achieved complete response and partial response to overall therapeutic intervention patients

CONTACTS AND LOCATIONS:
Overall Officials: Ming Gao, MD, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided